CLINICAL TRIAL: NCT07070206
Title: Effectiveness of Culturally Customised Maternal Nutrition Education for Health Professionals in Improving Their Counselling Capacity in Ethiopia
Brief Title: Culturally Customised Maternal Nutrition Education for Health Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahir Dar University (Other)
Responsible Party: Principal Investigator, Yeshalem Mulugeta Demilew, Associate professor, Bahir Dar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMHS, BDU; 2024 (Other Grant/Funding Number: Nestl Foundation); CMHS,BDU (Registry Identifier: Clinicaltrials.gov); BDU (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2025-01-28; First posted 2025-07-17 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Randomized Controlled Trial
Keywords: Counseling practice; Health professionals; In-service training

STUDY DESIGN:
Intervention Model Description: A two arm parallel cluster randomized controlled trial will be conducted in Bahir Dar city adminstration and Bahir Dar Zuria district, Ethiopia.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors willnot be aware about the objective of this intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- capacity building arm (Experimental): Health professionals in the capacity building arm will receive capacity building in-service training for the health professionals.
  Interventions: Behavioral: The health professionals in the capacity building arm will receive in-service training about culturally customized maternal nutrition education.
- routine capacity building arm (Other): Health professionals in the routine capacity building arm will receive capacity building in-service training given through the health care system.
  Interventions: Behavioral: The health professionals in the capacity building arm will receive in-service training about culturally customized maternal nutrition education.

INTERVENTIONS:
Behavioral: The health professionals in the capacity building arm will receive in-service training about culturally customized maternal nutrition education. — The health professionals in the routine capacity building arm will receive in-service training given through the health are system.
  Other Names: Routine capacity building in-service training

SUMMARY:
Background: Inadequate dietary consumption is a primary risk factor contributing to undernutrition during pregnancy and adversely affect birth outcomes. Despite this, in Ethiopia, 59.9% to 84.8% of pregnant women have inadequate dietary intake. Maternal nutrition education on healthy diet during pregnancy is one of the cost-effective interventions to improve dietary intake of pregnant women. However, nutrition education during pregnancy is not properly implemented in the country.

Objectives: The aim of this project is to investigate effectiveness of culturally customized maternal nutrition education for health professionals in improving their counseling capacity in Ethiopia.

Methods: A two arm parallel cluster randomized controlled trial will be conducted in Bahir Dar city adminstration and Bahir Dar Zuria district, Ethiopia, from 08/01/2024-8/20/2025. A Nonadjacent cluster (health institutions) will be selected using cluster sampling technique and randomized into the intervention and control groups. Data will be collected before and after the intervention using a structured questionnaire. Effect of the intervention will be assessed using generalized linear mixed-effects models.

Intervention strategies: The intervention will be in-service training about culturally customized maternal nutrition education for health professionals working at antenatal, delivery, and postnatal care units in the capacity building group. It will be given for five days monthly for four months using education guide. Health professionals in the routine capacity building group will receive routine capacity building training that will be given by the health system.

Project outcomes: Maternal nutrition counselling practices of health professionals will be the primary outcome.

DETAILED DESCRIPTION:
Introduction: Undernutrition during pregnancy is the main risk factor contributing to intrauterine growth retardation, premature delivery, low birth weight, and maternal and child mortality in Ethiopia. Despite this, the pooled prevalence of undernutrition in the country is 29%, ranging from 13.9% to 47.9%. Sub optimal dietary intake is the primary determinant contributing to undernutrition during pregnancy and it ranges from 59.9% to 84.8% in the country. Insufficient knowledge about healthy diet during pregnancy is the predictor for having inadequate dietary intake during pregnancy. Poor counselling practice of health professionals is a leading risk factor for poor maternal knowledge.

Nutrition education during pregnancy has a positive effect along the continuum from improving maternal knowledge about healthy diet to birth outcomes. According to a study in Dessie town, nutrition education improve nutritional knowledge scores of pregnant women from 6.9 to 13.4 and their dietary practices from 56.5% to 84.1%. Besides, nutrition education during pregnancy improve women's nutritional status and birth outcomes.

However, nutrition education during pregnancy is not properly implemented in the country. The current nutrition education practice is advising pregnant women to eat one additional meal from foods available at home compared to their preconception meals. This type of education is unclear for women since what is available at home is not specific and varies across households. Taking one extra meal may not be enough for all pregnant women, as nutrient requirements vary for different women and the trimester of pregnancy.

The bottlenecks for the current nutrition education are knowledge and skill gaps among health providers, limited nutrition education materials, and weak supportive supervision and feedback. This indicates the necessity of building health professionals capacity through nutrition education that takes into account communication and counselling skills. Since,in-service nutrition training for health professionals improve their knowledge and counselling practices. However, there is a paucity of evidence on the effectiveness of maternal nutrition education for health professionals in improving their counselling capacity in Ethiopia. Therefore, this study aims to investigate the effectiveness of in-service training about culturally customized maternal nutrition education for health professionals in improving their counselling capacity in Ethiopia.

This study will bring about a change in the current nutrition education implementation practice, health professionals' nutrition education competency, and generate evidence to guide maternal nutrition interventions. This project also has a long term benefit for maternal and child nutrition improvement.

Objectives

1 To estimate the effectiveness of culturally customized maternal nutrition education in improving health professionals' nutrition knowledge in Ethiopia, 2024 2. To estimate the effectiveness of maternal nutrition education in improving health professionals nutrition education practice in Ethiopia, 2024

Study setting and period: This study will be conducted in Bahir Dar city administration and Bahir Dar Zuria district, Ethiopia, from 08/01/2024-8/20/2025.

Study design: A two arm parallel cluster randomized controlled trial will be conducted in Bahir Dar City Adminstration and Bahir Dar Zuria district, Ethiopia.

Study population: The study population will be all health professionals who are working at antenatal, delivery, and postnatal care units in selected hospitals or health centers.

Sampling technique and sample size: Cluster sampling technique will be used to select the study participants, and health institutions will be considered as a cluster. First, nonadjucent clusters will be selected using simple random sampling (SRS) method. Then, 12 clusters will be selected after determining the required number of clusters using cluster size determination formula proposed by Rutterford C,et al, 2015.

Accordingly, to select equal health institutions from each district,14 non adjacent clusters (twelve health centers and two hospitals with nonadjacent catchment areas) will be selected using simple random sampling (SRS) method after preparing list of nonadjacent clusters as a sampling frame. Clusters will be randomized using a matched pair randomization technique. All health professionals working at antenatal, delivery, and postnatal care units of selected health institutions will be included in the study.

Intervention strategies: The intervention packages will be in-service training for health professionals working at antenatal, delivery, and postnatal care units. The training will be given about healthy diet during pregnancy. Additionally, culturally customized nutrition education materials will be given to the health professionals and supportive supervision will be done. .

The training modality will be interactive lectures, role plays, case scenarios, and practical sessions. The project team will prepare a training material by reviewing previous national and international guidelines and literature. The nutrition education materials will be guided by health behaviour change theories and models.

The contents of in-service training materials will be healthy diet using healthy eating plate and counselling and communication approach. It will include basics of maternal nutrition, components of healthy diet, portion sizes needed, frequency of meals, supplements, infection prevention measures, and behavioural theories and models. Project team members will provide training for the health professionals at the health institutions.

Five days training will be given monthly for four months. Each monthly training will consist of three sessions.Training modules, job aids, and leaflet with key messages will be given to all health professionals (trainees) to use and display in their antenatal and postnatal units. One week supportive supervision will be done after each training of health care providers in the intervention group to identify and solve any difficulties while implementing the training. Health professionals will counsel pregnant women for 30 minutes during giving each antenatal and postnatal cares. They will also educate pregnant and lactating women during monthly women's conference at the health institutions. They will counsel women using counselling guide with key points. The routine capacity building group will receive routine in-service training through the health system.

Data collection tools and procedures: Structured self administered questionnaire will be used to collect baseline data. Additionally, observational check lists will be used to assess counseling practices of health professionals. Three nurses will collect data and one supervisor will supervise data collection process.

Project outcomes: Counseling practice of health professionals will be the primary outcome while knowledge of health professionals will be the secondary outcomes. Birth weight will be tertiary outcome of this intervention.

Quality assurance mechanisms :Various measures will be taken to maintain the quality of the research, starting from designing the study to the data analysis and interpretation of the results. Fidelity of the intervention will be checked.

Data analysis strategies: The generalized linear mixed effects model will be used to analyze the effect of the intervention on health professionals' counseling practices. Health institutions will be analyzed as random effects in the regression model.

Ethical declarations: The Institutional Review Board of Bahir Dar University approved the study. Written consent will be secured from the study participants. The trial will be registered in the Clinical Trials.gov.

ELIGIBILITY:
Inclusion Criteria:Working in Antenatal, delivery and postnatal care clinics

-

Exclusion Criteria:

* On annual leave during enrolment of the study participants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Knowledge of the health professionals on diet during pregnancy will be the primary outcome of this study. | One year
  Health professionals' knowledge will be assessed using twenty four " yes/no " type questions on counselling and maternal diet. Health professionals who scored above 80% of knowledge assessment questions will be knowledgable, otherwise not knowledgeable.
Nutrition counselling practices of the health professionals will be the primary outcome of this study. | One year
  Counselling practices of health professionals will also be assessed using eighteen " yes/no " type questions that will be filled by observing health professionals nutrition counseling practices. Health professionals who properly practiced more than 80% practice related activities will have good counselling practice, otherwise not.

SECONDARY OUTCOMES:
Birth weight | one year
  Birth weight will be the secondary outcome of this intervention. Birth weight will be assessed using weighing scales.

CONTACTS AND LOCATIONS:
Overall Officials: Getu D Alene, Study Director — Bahir Dar University
Locations (1):
- Bahir Dar University, Bahir Dar, Amhara, Ethiopia

REFERENCES:
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Wakwoya EB, Belachew T, Girma T. Determinants of nutritional status among pregnant women in East Shoa zone, Central Ethiopia. Front Nutr. 2022 Dec 15;9:958591. doi: 10.3389/fnut.2022.958591. eCollection 2022. PMID 36590215
- [Background] Fite MB, Tura AK, Yadeta TA, Oljira L, Roba KT. Factors associated with undernutrition among pregnant women in Haramaya district, Eastern Ethiopia: A community-based study. PLoS One. 2023 Mar 9;18(3):e0282641. doi: 10.1371/journal.pone.0282641. eCollection 2023. PMID 36893154
- [Background] Demilew YM, Alene GD, Belachew T. Dietary practices and associated factors among pregnant women in West Gojjam Zone, Northwest Ethiopia. BMC Pregnancy Childbirth. 2020 Jan 6;20(1):18. doi: 10.1186/s12884-019-2702-z. PMID 31906981
- [Background] Demilew YM, Alene GD, Belachew T. Effect of guided counseling on dietary practices of pregnant women in West Gojjam Zone, Ethiopia. PLoS One. 2020 May 26;15(5):e0233429. doi: 10.1371/journal.pone.0233429. eCollection 2020. PMID 32453774